CLINICAL TRIAL: NCT05659615
Title: Applicability of New "Respiratory Diagnostic Assistant" Device in the Multidimensional Evaluation of Post-COVID-19 Respiratory Function
Brief Title: Analysis of Breathing Pattern Post COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shirley Lima Campos (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Universidade Federal de Pernambuco (Other)
Responsible Party: Sponsor-Investigator, Shirley Lima Campos, PhD, University of Pernambuco
Organization: University of Pernambuco (Other)
Other Study IDs: 44382120.3.0000.5208; 4.666.483 (Other: CEP-UFPE)
Record Dates: First submitted 2022-11-01; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Covid19
Keywords: COVID-19; Diagnosis; Physiotherapy; Breathing Pattern
MeSH Terms: conditions — COVID-19; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Study will not have intervention — Study will not have intervention

SUMMARY:
The COVID-19 pandemic, a disease caused by the SARS-CoV-2 virus, has generated an inexplicable scenario for global health, causing different complications and degrees of functional impairment in millions of people who manage to recover from the disease. The respiratory system is the main system to be directly impacted during COVID-19 infection, and its treatment can generate changes in the respiratory function of individuals surviving the exacerbation of the disease, which may promote subjective and quantitative changes in the respiratory pattern, requiring an evaluation with high-cost instruments, an evaluation necessary to outline a better planning therapeutic for this population. The goal of this study is evaluate the breathing pattern variables using a device called RESPIRATORY DIAGNOSTIC ASSISTANT (RDA) and verify the relationship between the breathing pattern variables with the variables of pulmonary function, respiratory muscle strength and respiration in patients after involvement by COVID-19. This is a observational and validation study, prospective with follow-up of respiratory function for 6 months, a subproject linked to the project already approved by the research ethics committee under opinion: 4.362.977/4.596.02. Data collection will be carried out in a single day and divided into a few steps that will take place at the cardiopulmonary physiotherapy laboratory located at the physiotherapy department of the Federal University of Pernambuco. The first step is to conduct an interview with the participants to collect clinical data and perform a physical examination. Subsequently, a multidimensional evaluation of respiratory function will be performed. Statistical analysis will be performed using the Statistical Package For Social Science (SPSS) software version 20.0 for Windows. The Kolmogorov-Smirnov test will be used to verify the type of distribution, regarding the normality of the variables, and the significance level adopted will be 95% (α <0.05) for all analyses. Finally, the data obtained will be presented in tables and/or graphs.

DETAILED DESCRIPTION:
The sample will consist of volunteers with laboratory confirmed COVID-19 results who have SARS COV 2 variants tracked by the epidemiological surveillance of Caruaru-Pernambuco and will be recruited by coexistence in a non-probabilistic way. The sample study will be obtained through data provided by the municipal health department of the city of Caruaru-Pernambuco with a predicted sample of 131 people. In order to minimize sample losses, 10% will be added to the total sample, which corresponds to 144 participants. The software that can be used is known as GPower (version 3.13 for Windows) considering a statistical power (β) of 80% and a significance level (α) of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years;
* Diagnosed with COVID-19;
* After the period of home isolation or hospital discharge;
* More than 40 days without the presence of symptoms associated with COVID-19;

Exclusion Criteria:

* Participants who are unable to perform the assessment tests or who present contraindications to the assessment of respiratory function;
* Those patients who prove reinfection by the new Coronavirus;
* Pregnant patients;
* Refusal to sign the Free and Informed Consent Form (FICF)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will consist of patients of both sexes, aged over 18 years, who had a confirmed diagnosis of the new coronavirus (COVID-19) through laboratory tests such as the molecular biology test (RT-PCR) or serological. This sample will be matched by 90 individuals according to sex and age group without a confirmed diagnosis of COVID-19 and with a self-report of absence of symptoms related to COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-20 (Estimated); Study Completion 2023-02-10 (Estimated)

PRIMARY OUTCOMES:
Breathing pattern diagnosis | "Until the Completion of the Study, On Average 1 Year"
  The algorithm of the "Respiratory Diagnostic Assistant" device relates the variables respiratory rate, tidal volume, minute volume, inspiratory flow, expiratory flow, relationship between inspiratory and expiratory times, providing classification of breathing pattern during rest breathing. The "Respiratory Diagnosis Assistant" algorithm provides through graphs allowing the classification of the diagnosis in normal or altered.
  * Normal breathing pattern described in frequency of cases. It is defined no changes by the algorithm of the "Respiratory Diagnostic Assistant".
  * Altered breathing pattern described in frequency of cases. It is defined by changing the breathing pattern variables captured by the flow sensor of the "Respiratory Diagnostic Assistant" device during breathing at rest.
Breathing pattern variables | "Until the Completion of the Study, On Average 1 Year"
  The algorithm of the "Respiratory Diagnostic Assistant" device relates the variables respiratory rate, tidal volume, minute volume, inspiratory flow, expiratory flow, relationship between inspiratory and expiratory times.
  The variables of the breathing pattern will also be quantitatively evaluated::
  * Respiratory rate in incursion per minute
  * Tidal volume (measured in liters)
  * Minute volume (measured in liters);
  * Inspiratory flow (measured in liters);
  * Expiratory flow (measured in liters);
  * Ti/Ttotal, (measured in segunds)
  * I:E , relationship between inspiratory and expiratory times
  * Volume vs time;
  * Flow vs time.

SECONDARY OUTCOMES:
Lung Function | "Until the Completion of the Study, On Average 1 Year"
  Lung function tests are usually performed with computerized systems that analyze the data and provide immediate results.
  The spirometer associates variables capable of tracing a functional diagnosis of the respiratory system:
  * Forced vital capacity (FVC) (measured in liters);
  * Forced expiratory volume in 1 second - (FEV1) (measured in liters);
  * Relationship between forced vital capacity (FVC) and
  * Forced expiratory volume in 1 second - (FEV1);
  Functional Diagnosis:
  * Normal
  * Obstructive ventilatory disorder (mild, moderate or severe)
  * Restrictive ventilatory disorder (mild, moderate or severe)
  * Mixed ventilatory disorder (with detection of obstructive and restrictive abnormality)
Assessment of lung volumes and capacities by ventilometry | "Until the Completion of the Study, On Average 1 Year"
  Non-invasive analogue assessment of lung volumes and capacities, easy to understand, with quantitative variables
  Respiratory rate (RR) (measured in incursion per minute) Minute volume (MV), (measured in liters) Tidal volume (TV), (measured in liters) Inspiratory capacity (IC) (measured in liters) Vital capacity (CL) (measured in liters)
Maximum inspiratory pressure (Manuvacuometry) | "Until the Completion of the Study, On Average 1 Year"
  Manuvacuometry: Non-invasive measurement of inspiratory muscle pressure.
  * Maximum inspiratory pressure (MIP measured in cmH2O)
  * Maximum predicted inspiratory pressure (MIP predicted %)
Maximum expiratory pressure (Manuvacuometry) | "Until the Completion of the Study, On Average 1 Year"
  Manuvacuometry: Non-invasive measurement of inspiratory muscle pressure.
  * Maximum expiratory pressure (MEP - cmH2O)
  * Maximum predicted expiratory pressure (MEP predicted %)

OTHER OUTCOMES:
Six-minute walk test | "Until the Completion of the Study, On Average 1 Year"
  Evaluation of functional capacity, through submaximal effort, through data obtained during a six-minute walk. The pre-test and post-test variables were measured:
  * BORG scale (scale from 0 to 10)
  * Perceived Effort (scale from 6 to 20)
  * Peripheral Oxygen Saturation (%)
  * Heart rate (measured in beats per minute)
  * Respiratory Rate (measured by breaths per minute)
  * Blood Pressure (mmHg)
  * Distance Traveled (measured in meters)
  * Expected Distance (%)
Palmar Grip Strength | "Until the Completion of the Study, On Average 1 Year"
  Assessment of handgrip strength through the dynamometry, measuring grip strength in a total of three repetitions, taking into account the greatest strength obtained in kilograms (kg/f)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley L Campos, Phd, Study Director — Universidade Federal de Pernambuco
Locations (1):
- Federal University of Pernambuco Department of Physiotherapy, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No
Não: Não há um plano para disponibilizar o IPD